CLINICAL TRIAL: NCT06608953
Title: A Prospective Randomized Controlled Trial of Effect of Enhanced External Counter Pulsation to Arterial Stiffness in Chronic Hemodialysis Patient
Acronym: EECP in HD
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Thana Thongsricome, MD (Other)
Responsible Party: Sponsor-Investigator, Thana Thongsricome, MD, Principal investigator, Chulalongkorn University
Organization: Chulalongkorn University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 246/62; TCTR20220202008 (Other: Thailand Clinical Trials Registry)
Record Dates: First submitted 2024-09-20; First posted 2024-09-23 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-09

CONDITIONS: Hemodialysis
Keywords: Enhanced external counterpulsation; Hemodialysis; Arterial stiffness; Pulse wave velocity; Central aortic blood pressure

STUDY DESIGN:
Intervention Model Description: Non sham-controlled, randomized study
Who Masked: Outcomes Assessor
Masking Description: Dana analysis personnels are blinded to the reaserch arms. The subjects are not blinded to the treatment (not sham-controlled).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Enhanced external counterpulsation (intervention) group (Experimental): Recieving enhanced external counterpulsation application during hemodialysis
  Interventions: Device: Enhanced external counterpulsation
- Controlled group (No Intervention): Recieve standard hemodialysis with optimal medical care

INTERVENTIONS:
Device: Enhanced external counterpulsation — A device applying external pneumatic cuff pressure to the lower limbs, thighs, and buttock sequentially in the diastolic phase synchronouslty with electrocardiography to assist the cardiac function via diastolic augmentation mechanism.
  Arms: Enhanced external counterpulsation (intervention) group

SUMMARY:
The objectives of this study are;

* To study effect of Enhanced External Counter Pulsation on arterial stiffness, as measured by pulse wave velocity, compared to standard hemodialysis treatment.
* To study effect of Enhanced External Counter Pulsation on central aortic blood pressure compared to standard hemodialysis treatment.
* To study effect of Enhanced External Counter Pulsation on cardiac index decline during hemodialysis compared to standard hemodialysis treatment.
* To study effect of Enhanced External Counter Pulsation on intradialytic hypotension events compared to standard hemodialysis treatment.
* To study effect of Enhanced External Counter Pulsation on blood biomarkers for endothelial dysfunction and vascular inflammation compared to standard hemodialysis treatment.
* To identify any adverse events from utilizing Enhanced External Counter Pulsation, such as pain or uncomfortable feeling, or even uncontrol hypertension.

ELIGIBILITY:
Inclusion criteria

* Patients aged 18 years old or older
* Patients received hemodialysis at King Chulalongkorn Memorial Hospital for at least 3 months
* Patients received hemodialysis frequency for at least 3 times/week with adequate hemodialysis, named single pool Kt/V of 1.2 or more, as calculated by Chula urea kinetic model
* Patients achieving proper dry weight, as determined by clinical assessment or by body composition monitoring (Fresineus company)

Exclusion criteria

* Patients with severe or unstable disease required emergent specific treatment such as severe infection or hemodynamic instability
* Patients with acute coronary syndrome within 1 month
* Patients received coronary artery bypass graft surgery or percutaneous transluminal coronary angioplasty within 3 months
* Patients with severe valvular heart disease and hypertrophic obstructive cardiomyopathy known before inclusion or detected by pre - allocation (within 12 months) echocardiographic assessment
* Patients with cardiac arrhythmia including atrial fibrillation or atrial flutter known before inclusion or detected by pre - allocation (within 12 months) 12 - lead electrocardiography
* Patients with known or suspected deep vein thrombosis or peripheral arterial disease
* Patients with thoracic aortic aneurysm detected pre - allocation (within 12 months) echocardiography or abdominal aortic aneurysm detected by pre - allocation (within 12 months) abdominal ultrasonography
* Patients with bleeding diathesis other than uremic bleeding, including anticoagulants use, but antiplatelets or local thrombolytics for vascular access stenosis/thrombosis are not included
* Patients with uncontrolled hypertension, defined as systolic blood pressure > 160 mmHg or diastolic blood pressure > 100 mmHg
* Patients with severe pulmonary hypertension known before inclusion or detected by pre - allocation (within 12 months) echocardiographic assessment
* Pregnant patients
* Patients who not willing to give a consent or who cannot legally give a consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Estimated)
Dates: Start 2020-02-13 (Actual); Primary Completion 2025-02-13 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Pulse wave velocity | Baseline, 1.5 months, and 3 months of research
  Pulse wave velocity is a well-proven marker of arterial stiffness.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Chulalongkorn University, Bangkok, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Thongsricome T, Kositanurit W, Siwamogsatham S, Tiranathanagul K. Enhanced external counterpulsation, focusing on its effect on kidney function, and utilization in patients with kidney diseases: a systematic review. Asian Biomed (Res Rev News). 2023 Oct 26;17(5):208-221. doi: 10.2478/abm-2023-0062. eCollection 2023 Oct. PMID 37899762